CLINICAL TRIAL: NCT04739826
Title: Evaluating Efficacy and Safety of Flumatinib Versus Nilotinib for Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia(CML-CP) : A Multicenter, Open-lable, Real World Study
Brief Title: Flumatinib Versus Nilotinib for Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: HS-2020-07SZ
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-07

CONDITIONS: CML, Chronic Phase; TKI
MeSH Terms: interventions — nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- flumatinib: flumatinib 600mg QD, fasting administration
  Interventions: Drug: Flumatinib Mesylate; Drug: Nilotinib Pill
- nilotinib: nilotinib 300mg BID, fasting administration
  Interventions: Drug: Flumatinib Mesylate; Drug: Nilotinib Pill

INTERVENTIONS:
Drug: Flumatinib Mesylate — Flumatinib mesylate tablets 600mg qd
Drug: Nilotinib Pill — Nilotinib Capsules 300mg bid

SUMMARY:
The ultimate goal of CML treatment is to improve survival, including overall survival (OS), progression-free survival (PFS), event-free survival (EFS), and treatment-free remission (TFR). TFR is a new therapeutic goal for chronic myeloid leukemia in chronic phase (CML-CP). In ENESTnd and DASISION trials, both nilotinib and dasatinib achieved DMR more effectively than imatinib. In the guidelines for diagnosis and treatment of chronic myeloid leukemia in China (2020 edition), flumatinib has been recommended as an appropriate first-line treatment for newly diagnosed chronic phase chronic myeloid leukemia (CML-CP) patients. There is no doubt that the second-generation TKIs show great advantages in deep molecular response, which further increases the possibility of achieving treatment-free remission. However, there is no direct comparative study to determine which TKI is better for de novo CML-CP. Thus, we conducted a multi-center, open-lable and real world study to compare the efficacy and safety between flumatinib and nilotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age;
2. CML-CP patients diagnosed with CML within half a year；Patients who have been using second-generation TKI nilotinib or flumatinib for first-line treatment in clinical practice, but the history of continuous treatment does not exceed 3 months；3.patients are allowed to receive hydroxyurea treatment before first-line treatment with nilotinib or flumartinib; patients treated with interferon for no more than 3 months and other TKIs for no more than 2 weeks;

4.Patients who must sign informed consent before screening

Exclusion Criteria:

1. T315I mutation ; Y253F/H, E255K/V, F359C/V/I mutations in the nilotinib group;
2. Entry into another therapeutic clinical trial;
3. Concomitant diseases that, according to the investigator's judgment, pose a serious risk to the patient's safety or completion of the study;
4. History of neurological or psychiatric disorders, including epilepsy or dementia;
5. Major surgery within 4 weeks prior to Day 1 of study;
6. Patients with another primary malignancy,unless the other primary malignancy is currently stable or does not need active intervention;
7. Women of reproductive age or men who are unable to use adequate methods of contraception, including women who are pregnant or breastfeeding;
8. ECOG≥3;
9. Patients who are unable to compliance with study or follow-up procedures;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed chronic-phase CML patients (CMP-CP) treated with flumatinib or Nilotinib
Sampling Method: Non-Probability Sample
Enrollment: 491 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Major molecular response rate at 12 months | 12 months
  Major molecular response is defined as ≤ 0.1% BCR-ABL/ABL% by international scale

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China